CLINICAL TRIAL: NCT00437593
Title: UHR-OCT and HD-OCT for Preretinal Membranes: Is There a Difference Between ICG and Membrane Blue? A Randomized Clinical Trial
Brief Title: UHR-OCT and HD-OCT for Preretinal Membranes: ICG Versus Membrane Blue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Binder Susanne, Univ. Prof. Dr, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FR-2-CI-2007
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2007-12

CONDITIONS: Retinal Diseases
Keywords: preretinal membrane; vitrectomy; uhr-oct; hd-oct
MeSH Terms: conditions — Retinal Diseases; Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ppVE, MP, ICG — surgery with ILM staining
Procedure: ppVE, MP, MB — Surgery with ERM staining

SUMMARY:
Using the UHR-OCT and HD-OCT to evaluate early postoperative changes in patients with diagnosis preretinal membrane after successfully performed pars-plana vitrectomy and membrane peeling with two different types of dyes.

DETAILED DESCRIPTION:
Surgical procedures performed are pars-plana vitrectomy and membrane peeling with or without cataract extraction and IOL implantation. The type of the dyes is randomized. The study is designed to include a total of tweny cases (10 cases with ICG and 10 cases with Membrane blue)

Main outcome measures are:

UHR-OCT, HD-OCT distance and near visual acuity and contrast sensitivity amsler grid secondary outcome measures are: OCT Stratus 3000 and visual field. Clinical examinations: preoperative, and follow-up examinations after 1 week, 1 months, 3 months, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Preretinal membrane
* Age between 18 and 85 years
* Combined surgery possible(phacoemulsification and vitreoretinal procedure)

Exclusion Criteria:

* Age-related macular degeneration
* Previous retinal detachment surgery
* Previous laser treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
UHR-OCT HD-OCT | 12 months
Distance Visual acuity | 12 months
Near Visual acuity | 12 months
Contrast sensitivtiy | 12 months

SECONDARY OUTCOMES:
OCT Stratus 3000 | 12 months
Visual Field | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Binder, MD, Study Chair — Ludwig Boltzmann Institue for Retinology and Biomicroscopic Lasersurgery
Locations (1):
- Rudolf Foundation Clinic, Vienna, Vienna, Austria